CLINICAL TRIAL: NCT04123184
Title: Oral Health Perception and Difficulties Encountered by Parents in the Implementation of Oral Hygiene of Children Under 6, Qualitative Study.-
Brief Title: Oral Health Perception and Difficulties Encountered by Parents in the Implementation of Oral Hygiene of Children Under 6
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0417
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Carious Disease
Keywords: Therapeutic patient education; Having one child who as less than 6 years old; Pediatric Dentistry; Oral Health; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A qualitative analysis was carried out on 15 participants, in 3 different places: the Montpellier health center, a pediatric odontology practice in Nîmes and a dentistry practice in Marseille.

Two methods of analysis were chosen: thematic analysis and word counting.

ELIGIBILITY:
Inclusion criteria:

Parent or caregiver with at least one child under 6 years of age, with Caod ≥ 1 and high RCI

Exclusion criteria:

* Patient refusing to participate in the study.
* Patient who does not understand the French language or who has difficulty expressing himself.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents or caregiver of the child, men or women, aged at least 18 years old, with a good understanding of the French language, accepting the terms of the study and not opposing its realization. The parent or caregiver with at least one child under the age of 6 who has a carious lesion or not.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the image that parents have of oral health and carious disease | 1 day
  Evaluation of the image that parents of oral health and carious disease by individual semi-guided interview

SECONDARY OUTCOMES:
Evaluation of the motivations and brakes encountered by parents in the implementation of oral hygiene of their child | 1 day
  Evaluation of the motivations and brakes encountered by parents in the implementation of oral hygiene of their child with early childhood caries (CPE) by individual semi-guided interview

CONTACTS AND LOCATIONS:
Overall Officials: Taormina Marion, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC